CLINICAL TRIAL: NCT02893202
Title: Examination of the Effects of Equine Assisted Activities [EAA] on Symptoms, Quality of Life and Functioning in Veterans With PTSD: An International Classification of Functioning, Disability and Health [ICF] Approach
Brief Title: Equine Assisted Activities on PTSD, Quality of Life and Functioning in Veterans With PTSD: An ICF Approach (THRICF)
Acronym: THRICF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: Horses and Humans Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EAAVeterans
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Equine assisted activities; quality of life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ride On Center for Kids (ROCK) facility (Experimental): 8-week therapeutic horseback riding
  Interventions: Other: Therapeutic Horseback riding
- Triple H Equitherapy Facility (Experimental): 8-week therapeutic horseback riding
  Interventions: Other: Therapeutic Horseback riding
- Rainer Therapeutic Riding facility (Experimental): 8-week therapeutic horseback riding
  Interventions: Other: Therapeutic Horseback riding
- REACH Therapeutic Riding facility (Experimental): 8-week therapeutic horseback riding
  Interventions: Other: Therapeutic Horseback riding
- Courtney Cares Riding facility (Experimental): 8-week therapeutic horseback riding
  Interventions: Other: Therapeutic Horseback riding

INTERVENTIONS:
Other: Therapeutic Horseback riding — An 8-week equine-assisted program designed to especially for veterans. The curriculum consists of eight 90-minute sessions designed to teach basic horse care and riding skills along with communication skills.

SUMMARY:
The purpose of the research project was to assess changes in Posttraumatic stress disorder [PTSD] symptoms, quality of life and participation of combat veteran who participate in equine assisted activities [EAA]. The study used a mixed-methods, waitlist-controlled, repeated measures trial of a standardized 8-week therapeutic riding intervention for combat veterans with PTSD. Behavioral changes were assessed four times during the study. Veterans meeting inclusion criteria were selected to participate in either the intervention group or the control/waitlist group.

DETAILED DESCRIPTION:
The research design was a quasi-experimental trial using mixed methods. Veterans recruited to a treatment group or a waitlist control group. Both qualitative and quantitative data was collected to assess changes. Qualitative data was collected post-intervention and quantitative data was collected at baseline, mid-intervention, post-intervention and 2-month follow-up.

A total of 125 veterans were recruited for the study. Eighty-nine met inclusion criteria.

Five therapeutic riding facilities will be utilized for this study: Ride On Center for Kids (R.O.C.K.), Georgetown, Texas; Riding Equines to Achieve Confidence and Health (R.E.A.C.H.), McGregor, Texas; Texas A&M Systems Courtney Grimshaw Fowler Equine Therapeutic Riding Center (Courtney Cares), College Station, Texas; Triple H, Cripple Creek, Texas, and Rainier Therapeutic Riding, Yelm, Washington. Two of the sites (R.O.C.K. and Rainier TR) are Professional Association of Therapeutic Horsemanship International [PATHIntl] premier accredited facilities, one (R.E.A.C.H.) is reaching premier status, and one (Courtney Cares) is under the direction of the research director at R.O.C.K. All four sites have existing Professional Association of Therapeutic Horsemanship [PATH] Equine for Service Members programs and the staff is experienced with the veteran population. Five sites were needed to ensure adequate sample size for the study.

EAA Protocol

The eight week EAA program followed the same protocol at all five testing sites with riding instructors and staff using a standardized curriculum, Rainier Therapeutic Riding's Riding Through Recovery. Baseline assessments was conducted for all participants in both the EAA group and the wait-list group. The EAA program consisted of eight, 90 minute weekly lessons. The first few lessons focused on developing a relationship between the horse and the participant without riding. The last two lessons included riding instruction if the participant chooses to ride. The PTSD Checklist- Military [PCL-M] and PTSD Checklist-5 [PCL-5] were administered pre and post as well as 2 months following the program. The Short Form Health Survey [SF-36v2], World Health Organization Disability Assessment Schedule 2.0 [WHODAS-2.0] and the Major Depression Inventory [MDI] were completed before beginning the program, at four weeks (mid-treatment), post-treatment and 2 months follow-up. Open-ended questions were completed post-treatment. The wait-list group participated in treatment as usual (TAU) and was assessed using the same instruments and time sequence with the exception of the post-treatment open-ended questions and the 2 month follow-up. After the first eight weeks, the wait-list group participated in the EAA intervention.

ELIGIBILITY:
Inclusion Criteria:

* participated in any of the three Iraq and Afghanistan war missions Operation Enduring Freedom, [OEF], Operation Iraqi Freedom,[OIF], Operation New Dawn, [OND]
* diagnosed with PTSD or exhibiting PTSD symptoms and confirmed using PCL-M or PCL-5 provisional diagnosis
* not participated in equine assisted activities and therapies six months prior to the start of the study

Exclusion Criteria:

* had a diagnosis of bipolar, schizophrenia, or presence of psychosis
* active substance dependence within the last three months
* significant cognitive impairment

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms | baseline, 4 weeks, 8 weeks, and 2 month post intervention
  PCL-5 to measure PTSD symptoms at each time point

SECONDARY OUTCOMES:
Change in behavior by participating in the program assessed with a semi-structured questionnaire | 8 weeks
  semi-structured questions designed to elicit responses about changes in behavior by participating in the program.
Change in Disability and Functioning | baseline, 4 weeks, 8 weeks, and 2 month post intervention
  WHODAS 2 was used to measure level of functioning at each time point
Change in Quality of life | baseline, 4 weeks, 8 weeks, and 2 month post intervention
  SF36v2 was used to measure quality of life at each time point
Change in Depression symptoms | baseline, 4 weeks, 8 weeks, and 2 month post intervention
  Major Depression Inventory was used to measure depression symptoms at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Lanning, PhD, Principal Investigator — Baylor University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ustun TB, Chatterji S, Kostanjsek N, Rehm J, Kennedy C, Epping-Jordan J, Saxena S, von Korff M, Pull C; WHO/NIH Joint Project. Developing the World Health Organization Disability Assessment Schedule 2.0. Bull World Health Organ. 2010 Nov 1;88(11):815-23. doi: 10.2471/BLT.09.067231. Epub 2010 May 20. PMID 21076562
- [Background] Ware, J. E., Kosinski, M., & Keller, S. D. (1994). SF-36 Physical and Mental Component Summary Measures: A User's Manual Boston: The Health Institute.
- [Background] Schneidert M, Hurst R, Miller J, Ustun B. The role of environment in the International Classification of Functioning, Disability and Health (ICF). Disabil Rehabil. 2003 Jun 3-17;25(11-12):588-95. doi: 10.1080/0963828031000137090. PMID 12959332